CLINICAL TRIAL: NCT02203175
Title: The Effect of Fentanyl-propofol Mixture on Propofol Injection Pain.
Brief Title: Prevention of Propofol Injection Pain
Acronym: VRS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, nurcan kizilcik, MD, Yeditepe University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 100-26.01.2011
Record Dates: First submitted 2014-06-30; First posted 2014-07-29 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: propofol; pretreatment; mixture
MeSH Terms: conditions — Pain | interventions — Sodium Chloride; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (plasebo): no pretreatment (Placebo Comparator): saline injection
  Interventions: Drug: saline; Drug: fentanyl; Drug: propofol
- propofol and fentanyl (Active Comparator): propofol 50 mg with fentanyl 50 mcgr iv during anesthesia induction ones time
  Interventions: Drug: fentanyl; Drug: propofol

INTERVENTIONS:
Drug: saline — Before the anesthesia induction, 5 ml isotonic saline
  Other Names: serum phisyologic
  Arms: Group C (plasebo): no pretreatment
Drug: fentanyl — before the anesthesia induction 50 mcgr fentanyl
  Other Names: talinat
Drug: propofol — during anesthesia 50 mg proposal with 50 mcgr fentanyl
  Other Names: pofol; diprivan

SUMMARY:
Pain on injection of propofol is a comman problem. The investigators planned to evaluate the effect of propofol-fentanyl mixture on propofol injection pain and compare it with fentanyl pretreatment and control groups.

Following ethics committee approval, 150 ASA I,II patients (18-65 yr) undergoing general anesthesia were enrolled to this study. Exclusion criteria were communication difficulty, psychiatric, neurologic disorders and history of allergy. Patients were randomly assigned to one of tree equal groups. Before the anesthesia induction, Group C (Control, n=50) and group M (mixture, n=50) received 5 ml isotonic saline, group F (fentanyl, n=50)received 2micgr/kg fentanyl. 10 seconds after the study drugs had been given, a standart question about the comfort of the injection was asked to the patient. The investigators used the verbal rating scale (VRS) for evaluation of propofol injection pain. Statistical analyses were performed with Student's t and Fisher's exact tests; p value <0,05 was considered significant.

Demographic data was similar among the groups (table I) In group M, the number of the patients having propofol injection pain was significantly lower compared to groups F and C (p<0,001 for both) None of the patients in groups F and M experienced severe pain whereas 24 patients (48%) had severe pain in group C (p<0.001 for both).

This study shown that fentanyl-propofol mixture is more effective compared to both fentanyl pretreatment and placebo in preventing propofol injection pain.

DETAILED DESCRIPTION:
150 ASA I-II patients, aged 18-65 year and scheduled for elective surgery were enrolled in the study. Patients were randomly assigned to one of three equal groups using an Excel (Microsoft , USA) generated randomization table. No patient received premedication. On arrival at the operation room after monitoring [ECG, noninvasive blood pressure, pulse oximeter and bispectral index (BIS)], a 20 gauge cannula was inserted into a vein on the dorsum of the patient's nondominant hand and %0.9 NaCl infusion was started at a rate of 5 ml/kg/h for 5 min, then i.v. infusion was stopped and the arm with the i.v. line was elevated for 15 s for drainage of venous blood. A tourniquet was placed on the forearm to produce a venous occlusion for 1 minute. The patients were pretreated by the anesthesiologist blinded to the groups. Before the anesthesia induction, Group C (Control, n=50) and group M (mixture, n=50) received 5 ml isotonic saline whereas group F (fentanyl, n=50)received 2micgr/kg fentanyl diluted with saline at a total volume of 5 ml as a pretreatment. (Propofol 1% Fresenius-FRESENIUS CABI- Fentanyl 0,05 mg/ml JANSSEN-CILAG ) The drugs were prepared by one of the investigators blinded to the study groups. Pretreatment solutions were identical in appearance. pH value of the fentanyl, propofol and fentanyl-propofol mixture was measured at the laboratory of our university with pH meter. For the patients in Group M a mixture of propofol and fentanyl was prepared using 20 ml propofol and 4 ml fentanyl. After the tourniquet was released, patients in Group C and F received 5 ml propofol whereas patients in Group M received 5 ml of this mixture. 10 seconds after the study drugs had been given, a standart question about the comfort of the injection was asked to the patient. We used the verbal rating scale (VRS) for evaluation of propofol injection pain. (0: none (negative response to questioning), 1: mild pain (pain reported only in response to questioning without any behavioral signs, 2: moderate pain (pain reported in response to questioning and accompanied by a behavioral sign or pain reported spontaneously without questioning), 3: severe pain (strong vocal response or response accompanied by facial grimacing, arm withdrawal or tears). All patients were able to answer the question about the pain and in all patients BIS was above 80 at that moment. The remaining dose of propofol and fentanyl was then given to complete the induction of anesthesia. Complete induction dose was propofol 2 mg/kg and fentanyl 2 mcg/kg. Because Group F and Group M had already received 2 mcg/kg fentanyl before, only Group C patients received 2mcg/kg fentanyl after the muscle relaxant. Before the induction of anesthesia, anesthesiologist explained all the patients that they will receive an iv. anesthetic that might lead to pain on the injection point, hand or arm.

STATISTICAL ANALYSES: Propofol injection pain was the primary outcome in the study. It is reported that the incidence of propofol injection pain is approximately 70 % and to decrease this incidence to 35% , it is calculated that 49 patients were needed in each group with a type I error of 0.05 and power of 90% . Due to possible drop outs in all groups 50 patients were taken into the study. Demographic data were compared with Student's t test . Fisher's Exact test and x2 tests were used to assess differences between categorical variables. A p value < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age
* ASA status I-II
* Scheduled for elective surgery

Exclusion Criteria:

* Communication difficulty
* Psychiatric and neurolojic disorders
* History of allergy to the study drugs
* Use of analgesics or sedative drugs within 24 hours before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
complete response | 1 year
  The primary outcome is complete response: A complete response is defined as no pain during proposal injection.

CONTACTS AND LOCATIONS:
Overall Officials: ferdi menda, assoc. prof., Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University Hospital, Istanbul, Devlet Yolu, Ankara Cad 102/104, Kozyatagi, Turkey (Türkiye)